CLINICAL TRIAL: NCT05239234
Title: Pre-operative Ultrasonographic Evaluation of Inferior Vena Cava Collapsibility Index and Caval Aorta Index to Predict Hypotension After Induction of General Anesthesia
Brief Title: Ultrasonographic Predictors of Hypotension After Induction
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: AntalyaTRH55
Record Dates: First submitted 2022-01-19; First posted 2022-02-14 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-01

CONDITIONS: General Anesthesia; Hypotension on Induction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Inferior vena cava-Aorta diameter index — Before the induction of general anesthesia, inferior vena cava-Aorta diameter index and inferior vena cava collapsibility index will be measured.
  Other Names: Inferior vena cava collapsibility index

SUMMARY:
The purpose of the study is to evaluate the predictive value of the inferior vena cava collapsibility index and caval aorta index for detecting hypotension after induction of general anesthesia.

DETAILED DESCRIPTION:
Since cardiovascular depressant and vasodilatory effects of anesthetic agents, patients may be at risk of hypotension after induction of general anesthesia. Previous studies reported that, for evaluating volume status, some ultrasonographic measurements such as inferior vena cava collapsibility index (IVCCI) could be used. Also some studies stated that measurement of aorta diameter index (IVC : Ao index) is reliable to predict hypotension after induction of spinal anesthesia. At the study, the investigators aimed to investigate the predictive values of the inferior vena cava collapsibility index and caval aorta index under ultrasound guidance in predicting post-induction hypotension in patients under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* patients more than 18 years of age
* American Society of Anesthesiologists' (ASA) physical status 1 or 2

Exclusion Criteria:

* BMI more than 30 kg/m²
* Use of angiotensin converting enzyme inhibitors
* pregnancy,
* emergency operations
* baseline arterial systolic blood pressure less than 90 mmHg
* mean arterial blood pressure less than 70 mmHg

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who scheduled for elective non-cardiac surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic value of IVCCI to detect post-induction hypotension assessed by Receiver operating characteristic (ROC) curve analysis. | 20 minutes
  Measurement of inferior vena cava collapsibility index.
Diagnostic value of IVC : Ao index to detect post-induction hypotension assessed by ROC curve analysis. | 20 minutes
  Measurement of inferior vena cava-Aorta diameter index.

CONTACTS AND LOCATIONS:
Overall Officials: Enes Eskin, M.D., Principal Investigator — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Researching Hospital, Antalya, Turkey (Türkiye)